CLINICAL TRIAL: NCT01516996
Title: Neoadjuvant and Concurrent Chemoradiotherapy Plus Nimotuzumab in Treating Patients With Locoregionally Advanced Squamous Cell Carcinoma of the Oropharynx and Hypopharynx
Brief Title: Safety and Efficacy Study of Nimotuzumab Plus Neoadjuvant and Concurrent Chemoradiotherapy to Treat Oropharynx and Hypopharynx Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second People's Hospital of Sichuan (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, LANG Jin-yi, Professor of radiotherapy department, The Second People's Hospital of Sichuan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-SCCHN-036
Record Dates: First submitted 2012-01-11; First posted 2012-01-25 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Oropharyngeal Cancer; Hypopharyngeal Cancer
Keywords: Neoadjuvant; Concurrent Chemoradiotherapy,CCRT; Nimotuzumab; Locoregionally Advanced Oropharynx; Hypopharynx cancer; Randomized; Multicenter
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Docetaxel; Cisplatin; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant and CCRT (Active Comparator)
  Interventions: Drug: docetaxel and cisplatin; Radiation: IMRT
- Neoadjuvant and CCRT and Nimotuzumab (Experimental)
  Interventions: Drug: docetaxel and cisplatin; Radiation: IMRT; Biological: Nimotuzumab

INTERVENTIONS:
Drug: docetaxel and cisplatin — * The neoadjuvant consists of docetaxel 75mg/m2 day 1 and cisplatin 75mg/m2 days 1 to 3, repeat every 3 weeks, for 2 cycles.
  * CCRT: cisplatin 75mg/m2 is administered on day 1 of week 7,10 and 13 on current with RT
Radiation: IMRT — IMRT is administered with chemotherapy from week 7 to week 13
  * GTV（primary tumor）：68-70Gy/35~38 F，once a day, 5 times per week
  * CTV（Clinical target）：56-66Gy/30~36f，once a day, 5 times per week
  * GTV-ln（positive neck region）：66-70Gy/33~36 F，once a day, 5 times per week
  * CTV-ln（negative neck region）：50-54Gy/28~30F, once a day, 5 times
  Other Names: CCRT
Biological: Nimotuzumab — Nimotuzumab was administered 200 mg IV over 1 hour on day 1,once a week, for 13~14 weeks
  Arms: Neoadjuvant and CCRT and Nimotuzumab

SUMMARY:
The purpose of this study is to evaluate the efficiency and safety of adding nimotuzumab to neoadjuvant and concurrent chemoradiotherapy in the treatment of patients with locoregionally advanced squamous cell carcinoma of the oropharynx and hypopharynx.

DETAILED DESCRIPTION:
Locoregionally advanced squamous cell carcinoma of the head and neck(LA-SCCHN) poses one of the most complex management challenges. This stage of disease is still potentially curable, but requires combined-modality therapy. Recent studies have showed that induction chemotherapy（neoadjuvant）reduced the 3-year distant relapse rate. Concurrent chemoradiotherapy(CCRT), on the other hand, has demonstrated a significant and consistent benefit in local control rates, but its impact on distant failure is inconsistent. Nimotuzumab is a novel EGFR-targeting monoclonal antibody that has the potential.to be used as a single agent or as a radio- and chemotherapy sensitizer for the treatment of SCCHN. Thus, investigators conducted a randomized, multicenter phaseⅡ study to compare the efficiency and safety of adding nimotuzumab to neoadjuvant and CCRT with neoadjuvant and CCRT in the treatment of patients with locoregionally advanced squamous cell carcinoma of the oropharynx and hypopharynx.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form
* Histologically confirmed locally advanced (stages III and IVb), squamous cell carcinoma of the oropharynx and hypopharynx
* The tumor mass had to be measurable
* Karnofsky performance status ≥70
* Life expectancy estimated than 6 months
* Hematologic: WBC≥4×109 /L , plateletes≥100×109 /L, haemoglobin ≥100 g/L；
* Hepatic: AST/ALT<1.5 times upper limit of normal (ULN)；serum bilirubin<1.5 times ULN;
* Renal: Creatinine<1.5 times ULN；

Exclusion Criteria:

* Known distant metastases
* Primary tumor and nodes received surgery(except of biopsy)
* Received other anti EGFR monoclonal antibody treatment
* Previous chemotherapy or radiotherapy
* Participation in other interventional clinical trials within 1 month
* Other malignant tumor (except of non-melanoma skin Cancer or carcinoma in situ of cervix)
* History of serious allergic or allergy
* History of Serious lung or heart disease
* Pregnancy or lactation women, or women with suspected pregnancy or men with willing to get pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months after all the treatment ending
  Objective Response Rate: Complete response (CR)+ partial response (PR) rates base on RECIST evaluation system.
The Number of Participants with Adverse Events | Participants will be followed during the treatment and 3 months after all the treatment ending ,an expected average of 26 weeks
  Record the Number of participants with adverse events and the Grades of the AE according to CTCAE v3.0 as the two measure of safety.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause,assessed up to 5 years
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Evaluate the Local control Rate in 1 to 5 years. | Participants will be followed every year for the duration of 5 years
  To evaluate each year until 5 years later
Tumor-Free Survival | From date of randomization until the date of first documented occurrence of primary, neck, distant relapse,assessed up to 5 years
Non-metastatic Rate | The time from randomization until distant relapse occur,assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi J Lang, M.D., Principal Investigator — Radiotherapy department
Locations (13):
- China (13):
  - Gansu Province Medical Science Institute, Lanzhou, Gansu
  - Guangxi Tumor Hospital, Nanning, Guangxi
  - GuiZhou Cancer Hospital, Guiyang, Guizhou
  - Neimenggu Tumor Hospital, Baotou, Neimenggu
  - The Tumor Affiliated Hospital of Ningxia Medical University General Hospita, Yinchuan, Ningxia
  - Qinghai Five Hospital, Xining, Qinghai
  - ShanXi Cancer Hospital, Xian, Shanxi
  - Xijing Hospital, Xi’an, Shanxi
  - The Second People's Hospital of Sichuan, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Sichuan
  - Xinjiang tumor hospital, The Third Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Tumor Hospital, The Third Affiliated Hospital of KUNMING Medical University, Kunming, Yunnan